CLINICAL TRIAL: NCT01802034
Title: Repository of Novel Analytes Leading to Autoimmune, Inflammatory and Diabetic Nephropathies (RENAL AID)
Acronym: RENAL AID
Status: Recruiting | Type: Observational
Sponsor: The Rogosin Institute (Other)
Collaborators: New York Presbyterian Hospital (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1207012648
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Kidney Diseases; Kidney Failure, Chronic; Diabetic Nephropathy; Lupus Nephritis; Glomerulonephritis, IGA
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Diabetic Nephropathies; Lupus Nephritis; Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, urine, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Native, Renal Tissue Preservation Group: Subjects who have a renal biopsy and the tissue is possessed and maintained by the RENAL AID repository.
- Native, Non-tissue Preservation Group: 1. Subjects who have had a renal biopsy but the tissue is not held by RENAL AID repository; and/or
  2. Subjects with diabetes and renal disease who have not had a renal biopsy.
- Transplant Nephropathy Group: Subjects who have had a renal transplant and require a transplant biopsy for either surveillance or "for-cause" indications.

SUMMARY:
A central goal of this data repository is to collect data from a large population of subjects with a variety of renal disease states. Cohorts will include subjects with diabetes, inflammatory/autoimmune and transplant related renal conditions. Additionally, the repository will have the capacity to store biospecimens and electronic data in control subjects without established renal disease. This initiative will provide an opportunity to compare data from various disease states and controls with the objective of determining clinical and biological factors that predict disease progression, response to therapy and identify discriminating noninvasive clinical and biological features that predict renal biopsy findings.

DETAILED DESCRIPTION:
RENAL AID is designed as an inclusive data and tissue repository that is capable of linking demographic, clinical, laboratory, histology, genetic and radiographic data into one interconnected electronic data collection instrument. It is hypothesized that by linking these typically disconnected data components into a single electronic repository, RENAL AID will be capable of discovering relationships between these otherwise disparate data sets in order to ascertain previously unknown factors and associations that contribute to the progression of disease, the incidence of complications (including renal failure) and response to therapy. Further, certain patterns of inflammatory and/or immune mediators present in the serum, whole blood and urine of subjects with renal disease may be predictive of the underlying histopathology present in renal biopsy specimens. The potential correlation of non-invasive markers with underlying histopathology in subjects undergoing renal biopsy may afford the ability to make renal diagnoses non-invasively in the future.

RENAL AID will obtain and follow clinical data on large numbers of subjects from a variety of ethnic, social and economic backgrounds in the following three research subject groups:

1. Native Biopsy Tissue Group: This group consists of subjects for which an expectant renal biopsy is undertaken based upon clinical necessity for whom surplus tissue is available. Subjects enrolled in this group will be evaluated every 3 months for the first year following biopsy, then annually thereafter. Research whole blood, serum and urine will be obtained at these visits.
2. Native kidney, non-tissue group: This group consists of subjects who have undergone a renal biopsy without specimen storage in the RENAL AID biorepository and/or subjects who have diabetes and concurrent kidney disease in the absence of a renal biopsy. Subjects enrolled in this group will be evaluated annually. Research whole blood, serum and urine will be obtained at these visits.
3. Allograft tissue group: This group consists of subjects that have undergone a renal transplant and require a transplant biopsy for either surveillance (termed protocol biopsy) or "for-cause" indications. By definition, "for-cause" biopsies are performed when an unexpected clinical event occurs that warrants transplant biopsy. Such events include acute graft dysfunction, progressive decline of transplant function, proteinuria and hematuria. Subjects in this group will be evaluated at the time of the transplant biopsy and research whole blood, serum and urine will be obtained at the visit.

Additionally, as RENAL AID is designed as both a biospecimen and data repository with the objective to conduct a wide variety of diverse research based upon the data and tissue collected, there will be research investigations for which control subjects are necessary. In anticipation of this requirement, RENAL AID will have the ability to record clinical, laboratory and histology data on control subjects in the same manner as for research subjects for those studies that obligate a control group and will have the ability to store bio-specimens and tissue in the same manner as for research subjects. In these circumstances, control subjects will be consented and RENAL AID will store electronic data and biopspecimens per protocol.

ELIGIBILITY:
Key Inclusion Criteria:

All Groups:

* Males or females
* 18 years of age and older
* Willing and able to provide informed consent

Native Biopsy Tissue Group:

- Require an initial kidney biopsy for medical necessity

Native Kidney, Non-tissue Group:

* Previously had a kidney biopsy and the tissue is not stored in this biorepository; or
* Have diabetes and kidney disease and have not had a kidney biopsy

Allograft Tissue Group:

- Have undergone a renal transplant and require a transplant biopsy for either surveillance or "for-cause" indications.

Key Exclusion Criteria for all Groups:

- Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from The Rogosin Institute, NewYork Presbyterian Hospital and affiliated institutions.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-02; Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in disease progression | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Perlman, M.D., Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States